CLINICAL TRIAL: NCT01841099
Title: Randomised Placebo-controlled Trial of a Gut Immunomodulatory Agent (Mesalamine) to Tackle Environmental Enteropathy in Acutely Malnourished Children: A Pilot Study.
Brief Title: Mesalamine in Environmental Enteropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kelsey Jones (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor-Investigator, Kelsey Jones, Study Principal Investigator, KEMRI-Wellcome Trust Collaborative Research Program
Organization: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KEMRI_CT_2013/0016; SSC 2223 (Other: KEMRI Scientific Steering Committee)
Record Dates: First submitted 2013-04-15; First posted 2013-04-26 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesalamine (Experimental): Mesalamine. Mesalamine granules. 30 mg/kg/day oral for 7 days followed by 50 mg/kg/day oral for 21 days if tolerated.
  Interventions: Drug: Mesalamine
- Placebo granules (Placebo Comparator): Placebo granules
  Interventions: Drug: Placebo granules

INTERVENTIONS:
Drug: Mesalamine — Mesalamine granules
  Other Names: Mesalazine, Pentasa (trade name)
  Arms: Mesalamine
Drug: Placebo granules — Provided by Ferring Pharma
  Arms: Placebo granules

SUMMARY:
Undernutrition is one of the most important health issues in Kenya. Children who are chronically undernourished do not reach their full potential and are at increased risk of infectious disease. Stunting occurs in a third of Kenyan children and has severe and long-term consequences in terms of health, development, and poverty. Several studies have shown that stunting is frequently associated with subclinical inflammation of the bowel, a condition referred to as Environmental Enteropathy (EE), previously known as 'tropical sprue' or 'tropical enteropathy'. EE is clinically similar to childhood inflammatory bowel diseases (IBD), including Crohn's disease. The treatment of IBD routinely involves provision of gut immunomodulatory agents, but this approach has never been tried in EE.

This proposal outlines a pilot double-blind randomised placebo-controlled trial of mesalamine (also called mesalazine - the safest immunomodulator used in IBD with least systemic activity) in treatment of severely malnourished children with EE.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 5 years old.
* Provision of informed consent by parent or guardian.
* Stunting (height for age z score <-2)
* Severe malnutrition (one or more of mid-upper arm circumference <11.5cm, weight for height z score <-3, or nutritional oedema).
* Eligible for outpatient management of malnutrition (i.e. no evidence of acute infection, and passes 'appetite test' according to national guidelines).
* Evidence of chronic inflammation (elevated erythrocyte sedimentation rate, ESR >20mm/hr).

Exclusion Criteria:

* Known HIV disease or tuberculosis.
* Known previous renal disease or asthma.
* Known allergy or hypersensitivity to mesalamine, other salicylate drugs, or any of the product ingredients.
* Biochemical evidence of acute renal or hepatic impairment on screening blood tests.
* Thrombocytopenia
* Recent (previous two weeks) bloody diarrhoea.
* Concurrent medication known to interact with the study drug (non-steroidal anti-inflammatory drugs, ranitidine, proton-pump inhibitors)
* Acute infection requiring treatment, e.g. lower respiratory tract infection or febrile illness.
* Other reason at the discretion of the attending clinician (independent of the trial team).

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events/serious adverse events | Day 0 to day 28 and day 0 to day 56
  This trial represents the first time a member of a class of drugs are to be used in a particular vulnerable group patient group. It's primary purpose is to conduct an early evaluation of safety and acceptability in this and the study is not powered to address any specific outcomes. It represents a modified Phase IIa design
Compliance with treatment | Day 0 to day 28
  This trial represents the first time a member of a class of drugs are to be used in a particular vulnerable group patient group. It's primary purpose is to conduct an early evaluation of safety and acceptability in this and the study is not powered to address any specific outcomes. It represents a modified Phase IIa design

SECONDARY OUTCOMES:
Changes in height | Day 0 to 28 and day 0 to day 56
  mm/day
Changes in levels of anti-Endotoxin Core IgG (EndoCAb) | Day 0 - Day 28 and Day 0 - Day 56
Changes in fecal calprotectin levels | Day 0 - Day 28 and Day 0 - Day 56
Changes in plasma soluble-CD14 | Day 0 - Day 28 and Day 0 - Day 56
Changes in plasma beta-2 microglobulin | Day 0 - Day 28 and Day 0 - Day 56
Changes in plasma neopterin | Day 0 - Day 28 and Day 0 - Day 56
Changes in weight | Day 0 - Day 28 and Day 0 - Day 56
  g/kg/day
Changes in mid-upper arm circumference | Day 0 - Day 28 and Day 0 - Day 56
  mm/day
Changes in C-Reactive Protein | Day 0 - Day 28, and Day 0 - Day56

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey DJ Jones, MBBS BA MRCPCH, Principal Investigator — KEMRI-Wellcome Trust Research Programme and Imperial College London
Locations (1):
- Baraka Clinic, Nairobi, Mathare, Kenya

REFERENCES:
- [Derived] Jones KD, Hunten-Kirsch B, Laving AM, Munyi CW, Ngari M, Mikusa J, Mulongo MM, Odera D, Nassir HS, Timbwa M, Owino M, Fegan G, Murch SH, Sullivan PB, Warner JO, Berkley JA. Mesalazine in the initial management of severely acutely malnourished children with environmental enteric dysfunction: a pilot randomized controlled trial. BMC Med. 2014 Aug 14;12:133. doi: 10.1186/s12916-014-0133-2. PMID 25189855